CLINICAL TRIAL: NCT03275805
Title: How Should Stable Graf Type IIc Hips be Treated With Pavlik Harness?
Brief Title: Should Graf IIc Hips be Treated for 12 Weeks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team determined that recruiting eligible patients is not feasible. Additionally, the PI retired in 01/2025.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-3104
Record Dates: First submitted 2016-11-21; First posted 2017-09-08 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Developmental Dysplasia of Hip
Keywords: DDH; Pavlik Harness; dysplasia
MeSH Terms: conditions — Hip Dislocation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12 weeks Pavlik Treatment Arm (Active Comparator): This arm will receive 12 weeks of full-time Pavlik Harness treatment. Patients will most likely begin the 12-week regiment at their first visit to our hip clinic.
  Interventions: Other: 12 week standard of care
- 6 weeks Pavlik Treatment Arm (Experimental): This arm will receive treatment to normalization, but for no less than 6 weeks. Patients will begin their treatment around the time of their first visit to our designated hip clinic.
  Interventions: Other: Duration of Pavlik Harness treatment

INTERVENTIONS:
Other: Duration of Pavlik Harness treatment — The only intervention that varies from standard of care (12 weeks of treatment) will be the duration of bracing (for the treatment to normalization arm). Patients in both arms will have identical follow up protocols and imaging to closely monitor hip morphology.
  Arms: 6 weeks Pavlik Treatment Arm
Other: 12 week standard of care — The intervention for this arm will be standard treatment for this pathology.
  Arms: 12 weeks Pavlik Treatment Arm

SUMMARY:
Children who are diagnosed with Developmental Hip Dysplasia (DDH) are often categorized depending on the severity of their hip malformation. Regardless of the severity, the accepted form of treatment is the Pavlik Harness. Unfortunately, there is no specific recommended treatment regarding length of Pavlik Harness treatment for patients with DDH who have who have been categorized with stable Graf type IIc hips. The investigators will aim to answer this question with a randomized controlled trial of patients with these specific findings by dividing selected patients into 2 arms. Each arm consists of varying lengths of Pavlik harness treatment (treatment to normalization, no less than 6 weeks or 12 weeks full-time). Patient's two year follow up radiographs will determine the best means of treatment.

DETAILED DESCRIPTION:
Developmental Dysplasia of the Hip is a thoroughly researched and manageable disease if treated correctly. While the literature agrees that Pavlik Harness treatment is the best means of treatment, there is still a lack of research regarding those patients who have stable Graf type IIc hips. Graf's classification method outlines the severity of dysplasia with a categorical method based on physical exam and ultrasound findings with a range of I-IV given in increasing order of severity. There are recommendations for how to treat more severe forms, but there is no consensus among orthopedic surgeons on how to specifically treat type IIc hips who present with stable hips.

Patients ages (0-18 weeks) of age will be recruited who present with stable Graf type IIc hips that have normal exam and abnormal ultrasound. The investigator's designated hip clinic defines normal exam as Ortolani and Barlow negative hips. Alpha angle will be used to determine normalcy on ultrasound. Abnormal ultrasound will be defined as an alpha angle <60 degrees, and less than 50% coverage and is justification in the facility for entrance into our designated hip protocol.

Upon meeting inclusion/exclusion criteria, patients diagnosed with IIc hips will be placed in the harness around 6 weeks of age. Patient consents will ensue at their 6 week follow up and will randomly divide patients into one of two arms: one control group which will receive the standard 12 week full-time protocol for Pavlik Harness treatment used at the institution, and one experimental group which will receive full-time Pavlik Harness treatment until normalization, but for no less than 6 weeks. All patients will be required to follow up at week 1, 2, 3, 4, 6, 8, 10, and 12, then at 6 months, one year, and two years from the time of harness placement. Ultrasounds will take place at week 1, 2, 3, 4, 6, 8, 10 and 12 and 6 months; radiographs will be taken at patients 6 month, one year and two year follow ups due to ossification of the femoral head. Acetabular Index (AI) at two-year radiographs will be used as the primary outcome variable.

Patients in the 6 week arm will only cease treatment if ultrasound and physical exam findings are acceptable. If patients fail to have acceptable ultrasound findings at 6 weeks, then the associated complication/failure will be noted, patients will be ineligible for study inclusion, and will continue with treatment to ensure hip reduction.

At routine follow ups, providers will note patient alpha angles on ultrasound at weeks 1,2,3,4,6, 8, 10, and 12 weeks. Since infant hips mature and may not be as visible on ultrasound around 6 months of age, acetabular indices on radiographs will be taken to measure patient hips at 6 month, 1 year, and 2 year follow ups. These images will be analyzed from within EPIC after patient visits and data information will be stored in RedCAP until the remainder of the study. Demographic and clinical characteristics will be included through descriptive statistics. Non-inferiority testing between patient's 2 year AI findings will determine if 6 weeks of treatment is no less harmful in terms of incidences of residual dysplasia to that of 12 weeks of treatment. The specified non-inferiority margin will be 4 degrees. This is the chosen clinically accepted difference in AI between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with:

* DDH
* Graf IIc hips (alpha angle = 43-49 degrees)
* normal hip exam (stable hips)
* abnormal ultrasound

Exclusion Criteria:

1. Patients with additional conditions: Neurologic or teratologic.
2. Follow up that occurs at any other institution.
3. Unstable hips

Ages: 0 Weeks to 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Acetabular Index at 2 years | 2 year follow up
  AI is a categorical measure that can be calculated on routine radiographs (X-rays). This measure helps clinicians get an overall view of the patient hip morphology and illustrates the effectiveness of Pavlik treatment by revealing the placement of the femoral head within the acetabulum (hip socket). AI is expressed as a horizontal line connecting Hilgenreiner's line to another line connecting the acetabular roofs.

OTHER OUTCOMES:
Cost of Treatment | After conclusion of the 2 year follow up
  Patient charges for both arms will be collected and compared (physician, imaging, facility charges)

CONTACTS AND LOCATIONS:
Overall Officials: Gaia Georgopoulos, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No sharing. Data is in RedCAP and will only be available for listed authors.

REFERENCES:
- [Background] Bialik V, Bialik GM, Blazer S, Sujov P, Wiener F, Berant M. Developmental dysplasia of the hip: a new approach to incidence. Pediatrics. 1999 Jan;103(1):93-9. doi: 10.1542/peds.103.1.93. PMID 9917445
- [Background] Dunn PM, Evans RE, Thearle MJ, Griffiths HE, Witherow PJ. Congenital dislocation of the hip: early and late diagnosis and management compared. Arch Dis Child. 1985 May;60(5):407-14. doi: 10.1136/adc.60.5.407. PMID 4015144
- [Background] Harding MG, Harcke HT, Bowen JR, Guille JT, Glutting J. Management of dislocated hips with Pavlik harness treatment and ultrasound monitoring. J Pediatr Orthop. 1997 Mar-Apr;17(2):189-98. doi: 10.1097/00004694-199703000-00010. PMID 9075094
- [Background] Herring JA. Conservative treatment of congenital dislocation of the hip in the newborn and infant. Clin Orthop Relat Res. 1992 Aug;(281):41-7. PMID 1499226
- [Background] Lorente Molto FJ, Gregori AM, Casas LM, Perales VM. Three-year prospective study of developmental dysplasia of the hip at birth: should all dislocated or dislocatable hips be treated? J Pediatr Orthop. 2002 Sep-Oct;22(5):613-21. PMID 12198463
- [Background] Mubarak S, Garfin S, Vance R, McKinnon B, Sutherland D. Pitfalls in the use of the Pavlik harness for treatment of congenital dysplasia, subluxation, and dislocation of the hip. J Bone Joint Surg Am. 1981 Oct;63(8):1239-48. PMID 7287794
- [Background] Novais EN, Sanders J, Kestel LA, Carry PM, Meyers ML. Graf Type-IV Hips Have a Higher Risk of Residual Acetabular Dysplasia at 1 Year of Age Following Successful Pavlik Harness Treatment for Developmental Hip Dysplasia. J Pediatr Orthop. 2018 Nov/Dec;38(10):498-502. doi: 10.1097/BPO.0000000000000875. PMID 27662383
- [Background] Paton RW, Hopgood PJ, Eccles K. Instability of the neonatal hip: the role of early or late splintage. Int Orthop. 2004 Oct;28(5):270-3. doi: 10.1007/s00264-004-0576-8. Epub 2004 Aug 12. PMID 15309324
- [Background] Rosendahl K, Dezateux C, Fosse KR, Aase H, Aukland SM, Reigstad H, Alsaker T, Moster D, Lie RT, Markestad T. Immediate treatment versus sonographic surveillance for mild hip dysplasia in newborns. Pediatrics. 2010 Jan;125(1):e9-16. doi: 10.1542/peds.2009-0357. Epub 2009 Dec 21. PMID 20026501
- [Background] Sewell MD, Rosendahl K, Eastwood DM. Developmental dysplasia of the hip. BMJ. 2009 Nov 24;339:b4454. doi: 10.1136/bmj.b4454. No abstract available. PMID 19934187
- [Background] Takahashi I. Functional treatment of congenital dislocation of the hip using Pavlik harness (Riemenbugel). Nihon Seikeigeka Gakkai Zasshi. 1985 Nov;59(11):973-84. PMID 3831166
- [Background] Westacott DJ, Mackay ND, Waton A, Webb MS, Henman P, Cooke SJ. Staged weaning versus immediate cessation of Pavlik harness treatment for developmental dysplasia of the hip. J Pediatr Orthop B. 2014 Mar;23(2):103-6. doi: 10.1097/BPB.0000000000000025. PMID 24322535
- [Background] Wood MK, Conboy V, Benson MK. Does early treatment by abduction splintage improve the development of dysplastic but stable neonatal hips? J Pediatr Orthop. 2000 May-Jun;20(3):302-5. PMID 10823594
- [Background] Atalar H, Sayli U, Yavuz OY, Uras I, Dogruel H. Indicators of successful use of the Pavlik harness in infants with developmental dysplasia of the hip. Int Orthop. 2007 Apr;31(2):145-50. doi: 10.1007/s00264-006-0097-8. Epub 2006 Apr 7. PMID 16601983
- [Background] Viere RG, Birch JG, Herring JA, Roach JW, Johnston CE. Use of the Pavlik harness in congenital dislocation of the hip. An analysis of failures of treatment. J Bone Joint Surg Am. 1990 Feb;72(2):238-44. PMID 2303510
- [Background] Lerman JA, Emans JB, Millis MB, Share J, Zurakowski D, Kasser JR. Early failure of Pavlik harness treatment for developmental hip dysplasia: clinical and ultrasound predictors. J Pediatr Orthop. 2001 May-Jun;21(3):348-53. PMID 11371819
- [Background] Graf R. Classification of hip joint dysplasia by means of sonography. Arch Orthop Trauma Surg (1978). 1984;102(4):248-55. doi: 10.1007/BF00436138. PMID 6712426
- [Background] Shorter D, Hong T, Osborn DA. Cochrane Review: Screening programmes for developmental dysplasia of the hip in newborn infants. Evid Based Child Health. 2013 Jan;8(1):11-54. doi: 10.1002/ebch.1891. PMID 23878122
- [Background] Woolacott NF, Puhan MA, Steurer J, Kleijnen J. Ultrasonography in screening for developmental dysplasia of the hip in newborns: systematic review. BMJ. 2005 Jun 18;330(7505):1413. doi: 10.1136/bmj.38450.646088.E0. Epub 2005 Jun 1. PMID 15930025
- [Background] Bracken J, Tran T, Ditchfield M. Developmental dysplasia of the hip: controversies and current concepts. J Paediatr Child Health. 2012 Nov;48(11):963-72; quiz 972-3. doi: 10.1111/j.1440-1754.2012.02601.x. PMID 23126391
- [Background] Shipman SA, Helfand M, Moyer VA, Yawn BP. Screening for developmental dysplasia of the hip: a systematic literature review for the US Preventive Services Task Force. Pediatrics. 2006 Mar;117(3):e557-76. doi: 10.1542/peds.2005-1597. PMID 16510634
- [Background] Patel H; Canadian Task Force on Preventive Health Care. Preventive health care, 2001 update: screening and management of developmental dysplasia of the hip in newborns. CMAJ. 2001 Jun 12;164(12):1669-77. PMID 11450209
- [Background] Godley DR. Assessment, diagnosis, and treatment of developmental dysplasia of the hip. JAAPA. 2013 Mar;26(3):54-8. doi: 10.1097/01720610-201303000-00011. No abstract available. PMID 23520807